CLINICAL TRIAL: NCT04490135
Title: Effectiveness of the Reitman Centre CARERS Group Intervention on Family Caregivers of Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Joel Sadavoy, Medical Director Reitman Centre, Mount Sinai Hospital, Canada
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARERSMountSinaiH
Record Dates: First submitted 2020-07-21; First posted 2020-07-28 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Carer Stress Syndrome
Keywords: Carer; Psychotherapy; Problem solving; Simulation; Dementia
MeSH Terms: conditions — Dementia | interventions — Psychotherapy, Group

STUDY DESIGN:
Intervention Model Description: a quasi-experimental design with a convenience sample and a non-randomized wait-list control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carers group intervention (Experimental): caregivers entered into the 8 week CARERS intervention (N=264) Group intervention, 8 x 2 hour sessions. Session 1-4 PST training, session 5-8 Simulation with standardized patients training Pre- post evaluations completed
  Interventions: Behavioral: Group psychotherapy
- Wating list control (No Intervention): Caregivers waiting for entry into active arm of CARERS intervention.During this time usual care allowed with no other intervention. Study measures administered at intake and immediately prior to starting the CARERS group. (N=83)

INTERVENTIONS:
Behavioral: Group psychotherapy — As described above
  Arms: Carers group intervention

SUMMARY:
Family caregivers (CG) of persons with dementia are vulnerable to disproportionate physical, mental and social adverse health consequences . The Reitman Centre CARERS program is an innovative, group psychotherapeutic skills-training intervention.

Study objective: to determine the effectiveness of the Reitman Centre CARERS program on key outcomes in family CGs of people with dementia. Study sample: Family CGs of people with dementia (n=264) referred to Reitman Center and the partner sites and wait-list control group (n=83) who received regular care. Method: quasi-experimental, non-randomized, multiple group trial; participants were evaluated before and after completion of the 8-week CARERS program in comparison.

DETAILED DESCRIPTION:
Addressing the adverse effects of caregiving on dementia CGs has been an increasing concern of mental and social health scholars in recent decades. Many single and multi-component programs have been developed but evidence for the effectiveness of interventions varies. Single component interventions for CGs like education, psychotherapy, or skills training are effective on various outcome measures but multicomponent programs appear to be preferred for overall reduction of caregiver burden. Broad development and system-wide adoption of interventions lags behind and there remains a need for evidence-based interventions that can be scaled widely in systems of dementia care.

This study aimed to compare the effectiveness of the Reitman Centre CARERS group intervention on measures of CG's health and well-being with a usual-care intervention control group. We hypothesized that the integrated, multicomponent CARERS program would produce robust positive effects on key outcome measures compared to waiting list controls. This was a quasi-experimental design with a convenience sample and a non-randomized wait-list control group implemented between 2013 and 2017. The control group received usual care before starting the CARERS intervention.The waiting list control group was derived from all CGs who were clinically assessed for the CARERS program, consented to enter the study and completed initial study assessments before being put on the waiting list for a CARERS group. A waiting list control was employed for practical recruitment purposes. This study was approved by the Sinai Health System (SHS) Research Ethics Board. Every participant provided informed signed written consent for all study components.Referrals to the study came from community agencies serving older adults, self-referrals, and primary care, memory, general psychiatry and geriatric medicine clinics. The intervention sites were located at Reitman Centre (CR) and Wellness Centre at Mount Sinai Hospital, Bridgepoint Active Health, Ceridian LifeWorks® EAP, Canadian Alzheimer Society chapters and community agencies serving older adults.

The intervention, called Carers, is a multicomponent, group psychotherapeutic, skills-training intervention for family CGs comprised of 8 weekly 2 hour closed groups sessions. of 4-6 CGs co-led by 2 mental health clinicians who follow a protocol that includes predetermined agendas that structure the outline of each group. The group leaders are trained to elicit and address the specific concerns of each CG during each session. The content of each group is determined by the CGs based on an initial go-round check-in to elicit current caregiving problems and challenges, emotional reactions and foster group cohesion. In sessions 1-4, CGs are formally taught a form of problem-solving therapy (PST) adapted for dementia CGs. Sessions 5-8 utilize simulation to train CGs to effectively communicate with the person they are caring for and learn how to engage with them to manage dementia induced behaviours such as resistance or demandingness. Communication training is done with live therapeutic simulation a hands-on training method that employs specially trained standardized patients (SP) in a tightly controlled intervention developed for the CARERS program. All group leaders were trained in a standardized training protocol at the Reitman Centre. CGs completed self-administered questionnaires at entry to the study, just prior to starting the first group and, immediately after session 8 of the group therapy. Care recipient (CR)function and demographic and socioeconomic information was gathered for each CG/CR at entry into the study. Statistical analysis employed IBM SPSS 26 and univariate general linear model (UNIANOVA) analysis and parametric tests.

ELIGIBILITY:
Inclusion Criteria:

* adult, informal caregiver (CG) of a person with diagnosis of dementia who resided in the community; sufficient emotional and physical capacity to participate in the assessment and training sessions; no active suicidality or psychotic illness; willing to discontinue other CG intervention programs while in the study; and provided signed consent for the study.

Exclusion Criteria:

* insufficient emotional and physical capacity to participate in the assessment and training sessions; active suicidality or psychotic illness; unwilling to discontinue other CG intervention programs while in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale- CESD) Eaton et al., 1977 | Change in depression score from baseline at 8 weeks
  standardized diagnostic measure of depression
perceived stress scale - PSS Cohen, S et al., 1983 | Change in stress score from baseline at 8 weeks
  self assessment standardized measure of self perceived stress
Mastery (Pearlin et al., 1990) | Change in mastery score from baseline 8 weeks
  self assessment standardized measure of perceived sense of mastery in caregiving
caregiving competence(Pearlin et al., 1990) | Change in caregiving competence score from baseline at 8 weeks
  Self assessment standardized measure of key areas of perceived competence in caregiving
role captivity (Pearlin et al., 1990) | Change in role captivity score from baseline at 8 weeks
  Self administered standardized measure of degree of perceived entrapment in the caregiving role
role overload(Pearlin et al., 1990) | Change in role overload score from baseline at 8 weeks
  self administered standardized measure of degree of experienced caregiving overload
Short Zarit Burden Inventory- SZBI), (Bedard et al., 2001) | Change in burden score from baseline at 8 weeks
  Self administered Standardized measure of burden of caregiving
coping (Endler and Parker 1990) | Change from Baseline at 8 weeks
  Self administered scale of caregiver's perception of coping
coping (Endler & Parker, 1990) | Change in coping from baseline at 8 weeks
  Self administered scale of caregivers perception of coping

SECONDARY OUTCOMES:
Caregiver demographics | through study completion on average about 4 months
  general demographic profile
Katz Index of Independence in Activities of Daily Living (Katz ADL) (Katz, Downs, Cash, & Grotz, 1970) | change from Baseline at 8 weeks
  Measure of care recipient daily function as observed by caregiver
Lawton Instrumental Activities of Daily Living Scale (Lawton ADL) (Lawton & Brody, 1969) | Change from Baseline at 8 weeks
  measure of care recipients daily instrumental activities of daily living as observed by the caregiver
Revised Memory and Behaviour Checklist- RMBPC) (Teri et al., 1992) | Baseline and after completion of the 8 week intervention
  Caregiver's reaction to CR's memory and behavioural symptoms (completed by caregiver)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Sadavoy, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Joel Sadavoy, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No